# Statistical Analysis Plan (SAP)

Sweet Tooth: Nature or Nurture? Role of Long-term Dietary Sweetness Exposure on Sweetness Preferences

Version 2024.02.07 (yyyy.mm.dd)

| GENERAL INFORMATION | |
|---|---|
| Principal investigator | Dr. M (Monica) Mars |
| | Sensory Science and Eating Behaviour |
| | Wageningen University and Research |
| | Wageningen, the Netherlands |
| | Dr. Kees de Graaf (Project leader) <sup>1</sup> |
| | Dr. João Paulo (statistician) <sup>1</sup> |
| | Dr. Katherine Appleton <sup>2</sup> |
| | Eva Marija Čad <sup>1</sup> |
| | Claudia Tang <sup>2</sup> |
| | Leoné Pretorius <sup>2</sup> |
| Core team members | Hanne de Jong <sup>1</sup> |
| | <sup>1</sup> Division of Human Nutrition and Health, Wageningen University and |
| | Research, Wageningen, The Netherlands |
| | <sup>2</sup> Department of Psychology, Faculty of Science and Technology, |
| | Bournemouth University, Bournemouth, United Kingdom |
| Name of project | Sweet Tooth |
| ClinicalTrials.gov identifier | NCT04497974 |
| Project Registration number | NL72134.081.19 |
| Ethical review | METC-nr 20/02, METC-WU |

# INTRODUCTION

**Primary objective:** To assess the effect of a 6-month low, regular, and high dietary sweetness exposure on preference for sweet foods and beverages, and to compare these effects between the intervention groups.

# **Objectives**

**Secondary Objective(s)**: To assess the effect of a 6-month low, regular, and high dietary sweetness expo- sure on taste intensity perception, behavioural outcomes: food choice and intake, sweet-liker type, food cravings, dietary taste preferences, dietary taste patterns; anthropometric outcomes: body composition, waist-hip circumference, body weight; and biochemical outcomes: glucose variability, and biomarkers related to CVD and diabetes.

| STUDY METHODS | |
|---|---|
| | The Sweet Tooth study is a 6-month parallel randomized controlled trial with partial food |
| Trial design | provision. with three arms: |
| | 1. a regular sweet exposure diet (RSE, control) (n=60); |
| | 2. a low sweetness exposure diet (LSE) (n=60); and |
| | 3. a high sweetness exposure diet (HSE) (n=60). |
| | Data collected at the screening visit are used to assign participants to intervention groups. |
| | Matched groups are randomized to the interventions to minimize differences between |
| | intervention groups in these baseline characteristics. Based on sex (2 levels: male, female), |
| Randomization | age (3 levels: 18-34, 35-49, 50-65), Body Mass Index (BMI) (2 levels: 18.5-24.9, 25-30 kg/ |
| | m2) and sweet liker phenotype (3 levels: sweet liker, inverted U, sweet disliker), in a process |
| | of stratified randomization (2×3x2×3=36 strata). Treatment allocation is performed |
| | according to a computer-generated random schedule, at the ratio 1:1:1 to each of the three |
| | groups. Treatment allocation is performed by an independent person, not involved in the |
| | study outcome assessments or statistical analyses. |
| | The sample size calculation is based on our primary outcome: change in preference score |
| | from 0–6 months. Previous studies have established that it is possible to detect shifts in |
| | preferred concentration from preference tests. For example, looking at the study of Liem |
| | and de Graaf (2004) and the change in most preferred concentration, we can observe that |
| Samuela sias | mean ranking score for the sweet exposure group changed by around 0.4 and by around |
| Sample size | 0.6 for the sour exposure group from baseline to after exposure, which is around 10%. |
| | Therefore, the effect size of 0.1 was considered to be a relevant and meaningful effect size |
| | for our study and was used to estimate the sample size. We estimate that 147 participants |
| | are needed to detect an effect size of 0.1, assuming a parallel study with 3 groups, with two |
| | repeated measures (baseline vs 6-month, correlation between measures of 0.7), and a |

| interim analysis<br>Timing of final | | - | | | | No interim analyses will be carried out. | | | |
|---|---|---|---|---|---|---|---|---|---|
| Timing of final | | | | | | | | | |
| Timing of final | Ctatistical analys | مأسم مما النبيية | rmand whan the | lost su | bioet I | | ba falla | | |
| - | Statistical analys | sis will be perio | imed when the | iast su | bject i | eaves t | ne rond | ow up p | period. |
| analysis | | | | | | | | | |
| | Domain | Outcome to Be | Data Collection | Baseline | Intervention | | | Follow-up | |
| | | Measured | Method | | 1Month | 3 Months | 6 Months | 7 Months | 10 Months |
| | Food taste preference | Sweetness preferences | Rank-rating scale | / | / | / | / | / | / |
| | r ood taste preference | Saltiness preferences | name racing scare | / | / | / | / | / | / |
| | Taste intensity percep- | Sweet taste perception | 100-unit VAS | / | / | / | / | / | / |
| | tion | Salt taste perception | | / | 1 | / | 1 | / | / |
| | Behavioural outcomes | Food choice | Food choice from a<br>buffet | 1 | 1 | ✓ | 1 | 1 | 1 |
| | | Food intake | Amount consumed from<br>a buffet | 1 | 1 | 1 | ✓ | 1 | 1 |
| | | Sweet-liker type | 100-point VAS | / | 1 | / | 1 | / | / |
| | | Taste preferences | PrefQuest <sup>a</sup> | ✓ | / | / | ✓ | ✓ | ✓ |
| | | Food cravings | CoEQ | / | 1 | / | 1 | ✓ | ✓ |
| Timing of | | Dietary taste patterns | Taste FFQ <sup>b</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| outcome | Anthropometric out- | Body composition | DEXA | ✓ | | | 1 | | 1 |
| outcome | comes | Waist-hip circumference | Measuring tape | / | / | / | / | / | / |
| assessments | | Weight | Digital scale | / | / | <b>✓</b> | / | <b>✓</b> | <b>✓</b> |
| | Biochemical outcomes | Biomarkers related to<br>CVD and diabetes | Fasting blood sample | / | / | / | / | / | / |
| | | Glucose homeostasis | Glucose sensor <sup>c</sup> | / | | | / | | / |
| | Compliance | Biomarkers of compli-<br>ance | Urine sample (24-h<br>sample) | 1 | / | 1 | 1 | 1 | 1 |
| | | Dietary intake | Online 24-h recall | / | / | / | / | / | / |
| | Intervention Modera- | Physical activity | SQUASH | ✓ | 1 | ✓ | ✓ | ✓ | ✓ |
| | tors | Adverse events, medica-<br>tion use | Questionnaires <sup>b</sup> , Study<br>diet diary | / | / | / | ✓ | / | ✓ |

| OUTCOMES | | |
|---|---|---|
| Primary Outcome measure | | |
| Outcome Measure | Measure Description | Time Frame |
| Change in preference score | Measured during preference testing, using Ranking on a scale methodology (scale anchored at 0: Dislike extremely; 50: Neither dislike or like; 100: Like extremely) in a series of test foods. | From month 0 to month 6. |
| Secondary Outcome measu | ires | |
| Outcome Measure | Measure Description | Time Frame |
| Change in preference score. | Measured during preference testing, using Ranking on a scale methodology (scale anchored at 0: Dislike extremely; 50: Neither dislike or like; 100: Like extremely) in a series of test foods. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Difference in mean liking scores between familiar and unfamiliar foods. | Measured during preference testing, using Ranking on a scale methodology (scale anchored at 0: Dislike extremely; 50: Neither dislike or like; 100: Like extremely) in a series of test foods. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Change in sensory intensity scores. | Measured during sensory testing, using 100-unit Visual analogue scale (VAS), (anchored at 0: not sweet/salty at all; 100: Extremely sweet/salty) in a series of test foods. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Change in energy intake. | Measured during ad-libitum test meal in kcal. | Measured at 0, 1, 3, 6, 7 and 10 months. |

| Change in energy intake. | Measured during ad-libitum test meal in kJ. | Measured at 0, 1, 3, 6, 7 and 10 months. |
|---|---|---|
| Proportion of eaten sweet foods vs. foods from other taste modalities. | Measured during ad-libitum test meal in proportions. | Measured at 0, 1, 3, 6, 7 and 10 months |
| Sweet-liker status score. | Measured on a 100-unit VAS scale (anchored at 0: Dislike; 100: Like). | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Food craving questionnaire scores. | Measured using the Control of eating questionnaire (CoEQ) | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Taste preference questionnaire scores. | Measured using Taste Preference questionnaire (PrefQuest). | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Dietary taste patterns. | Measured with the Taste food frequency questionnaire in frequency. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Dietary taste patterns. | Measured with the Taste food frequency questionnaire in % of energy coming from each taste cluster. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Dietary taste patterns. | Measured with the Taste food frequency questionnaire in % of food weight coming from each taste cluster. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Body weight. | Measured with a weighing scale in kg. | Measured at 0, 1, 2, 3, 4, 5, 6, 7 and 10 months. |
| Waist-to-hip ratio. | Measured using a stretch-resistant tape. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| % of body fat mass and lean body mass (fat free mass). | Measured with a dual energy x-ray absorptiometry (DEXA). | Measured at 0, 6 and 10 months. |
| Variation in interstitial glucose levels. | Measured with glucose monitoring sensor (only measured in a subgroup, of 60 subjects, 20 per intervention arm). | Measured at 0, 6 and 10 months. |
| Change in fasting glucose,<br>HbA1c, insulin, total<br>cholesterol, low-density<br>lipoprotein (LDL), high-<br>density lipoprotein (HDL),<br>triglycerides levels in<br>blood. | Measured in blood in mmol/L. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Concentration of biomarkers in urine related to sugar, low and no calorie sweeteners, protein and salt intake. | Measured in urine in mg/d. | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Intake levels of foods, food groups and macronutrients. | Measured with 24-hour recalls, in kcal/day. | Measured at 0, 1, 2, 3, 4, 5, 6, 7 and 10 months. |
| Other Outcome measures | | |
| Outcome Measure | Measure Description | Time Frame |
| Adverse events. | Self-reported and monitored. | Measured at 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months. |
| Gender. | Self-reported. | Assessed at month 0. |
| Height. | Measured with a stadiometer. | Assessed at month 0. |
| Physical activity level. | Measured with the Short Questionnaire to Assess<br>Health enhancing physical activity (SQUASH). | Measured at 0, 1, 3, 6, 7 and 10 months. |
| Polymorphisms related to sweet taste perception. | Genes will be extracted from collected blood samples. | Assessed at month 0. |
| Age. | Self-reported. | Assessed at month 0. |
| Medicine usage. | Number and type of medicine used, self-reported. | Assessed at month 0. |

| STATISTICAL PRINCIPALS | |
|---|---|
| Principals and P-<br>values | Prior to data analysis, normality of the data will be inspected. Non-normally distributed |
| | data will be transformed or analysed using non-parametric tests, if deemed necessary. |
| | Statistical significance is set at p<0.05. |
| Adherence and | Adherence to diets will be assessed on group level with biomarkers of sweetener |
| Protocol deviations | consumption in 24-h urine sample, and 24h recalls. |

#### STATISTICAL ANALYSIS

### **Analysis methods**

Data will be analyzed in R. Based on findings of previous studies (Liem and de Graaf, 2004), we do not expect the data to be non-normally distributed. Descriptive statistics will be provided for each of the three intervention groups at baseline and will include demographic, dietary and lifestyle information. Continuous data will be summarized using means, SD/SE and 95% confidence intervals or median/geometric means and backtransformed 95% Cl's if not normally distributed. Categorical variables will be summarized using counts and percentages.

Analysis will be conducted on both an intention-to- treat (ITT) and a per-protocol basis. The ITT analysis will be the primary analysis. The per-protocol analysis (participants who finished the study), will help us determine whether the effects are the result of individuals adhering to the procedure and consuming the provided intervention foods. In the event of missing data due to drop-out, the outcome variables that have not been recorded will be treated as missing data. Unblinding will occur at the conclusion of the study to determine the effect of the intervention. Unblinding will take place in two steps: initially disclosing the allocation of individuals to their respective groups, without indicating intervention allocation. Only after the primary analyses have been conducted we will unblind the identity of each group.

## **Primary outcome:**

To determine whether there is a shift in sweetness preference between baseline and month 6, statistical techniques appropriate for longitudinal data analysis, that is linear mixed effects models, will be used, with treatment (LSE, RSE and HSE), time (baseline, 1, 3, 6, 7 and 10-months) as fixed factors, the interaction between treatment x time outcome and participant number as a random factor. Our main interest is in the change in preference score between 0 and 6 months of any two intervention groups. The interaction effect will be evaluated to indicate if the change differed between the groups. If significant, the following predefined contrasts will be calculated: baseline vs. month 6 and LSE vs. RSE vs. HSE with all possible combinations. Subsequent, pairwise post-hoc tests will be Bonferroni adjusted.

#### Other outcomes:

Similar linear mixed effects models will be used to explore effects of sweet taste exposure on the other dependent measures over time (baseline, 1, 3, 6, 7 and 10-months). The interaction effect (intervention group x time) will be evaluated to indicate if the pattern of change of a certain outcome differed between the groups. If significant, the following predefined contrasts will be calculated: baseline vs. 1 vs. 3 vs. 6 vs. 7 vs. 10-months and LSE vs. RSE vs. HSE with all possible combinations.

In light of the research in this area, we will explore differences between intervention groups and secondary outcome variables and explore related but separate questions of whether glucose variability, body composition, food cravings, blood biomarkers are related to sweetness exposure, age, gender, sweet liker status and BMI.

By comparing group means of urine extraction of urinary sucrose, fructose, and LCSs between intervention groups, the level of compliance will be evaluated. Linear mixed effects models will be adjusted for covariates where appropriate and both unadjusted and adjusted models will be reported. If interaction effect between time and intervention are identified, Posthoc tests (with Bonferroni adjustments) will be applied to identify statistically significant differences.